CLINICAL TRIAL: NCT05782686
Title: Reduction of Affected Margins in Conservative Surgery for Breast Cancer: Impact of Systematic Shaving in the Operating Room
Brief Title: Impact of Systematic Shaving on Margins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, Clinical Professor, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR275/20
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Margin, Tumor-Free; Breast Cancer; Surgery
MeSH Terms: conditions — Margins of Excision; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed by another investigator outside the operating room after lumpectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shaving (Experimental): Subsequent to lumpectomy, a circumferential enlargement of all lumpectomy margins, including lateral, medial, superior, inferior, anterior, and posterior, approximately 5-10mm thick, will be resected.
  Interventions: Procedure: Margin shaving
- No Shaving (Active Comparator): Standard lumpectomy
  Interventions: Procedure: Margin shaving

INTERVENTIONS:
Procedure: Margin shaving — In both cohorts, an intraoperative study of the margins will be carried out, and enlargement of those margins that are affected will be carried out as indicated by the pathologist. Subsequently, shaving is performed in case of being randomized to the study group or surgery is completed in the control group.

SUMMARY:
The objective of this clinical trial is to demonstrate the reduction of positive margins in the definitive pathology of patients undergoing breast-conserving surgery with the systematic shaving technique compared to conventional surgery, and the reduction of second interventions for margin enlargement.

DETAILED DESCRIPTION:
Patients with breast cancer who undergo breast-conserving surgery are randomized in the operating room after lumpectomy into 2 groups of 117 patients each: shaving/no-shaving (standard surgery).

ELIGIBILITY:
Inclusion Criteria:

1. Breast-conserving surgery.
2. Imaging diagnosis as the only breast tumor focus according to mammography, breast ultrasound and/or nuclear magnetic resonance;
3. Pathological diagnosis of carcinoma in situ or infiltrating
4. Oncoplastic without associated flaps;

Exclusion Criteria:

1. Male patients;
2. Patients with a history of ipsilateral breast cancer.
3. Oncoplastic that includes flaps
4. Multifocality or multicentricity;
5. Pregnant or lactating patient;
6. Stage IV patients;
7. Patients eligible for mastectomy;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Margin involvement | 3 weeks after each surgery
  To compare the number of cases with affected margins in the definitive pathological anatomy, of the cases with intraoperative systematic shaving versus the group of no shaving
Re-interventions | 3 weeks after each surgery
  Demonstrate the reduction of second surgeries to widen affected margins in breast conserving surgery with the shaving technique

SECONDARY OUTCOMES:
Shaving versus intraoperative pathological study | 3 weeks after each surgery
  Assess the possibility of replacing the intraoperative study of the margins with systematic shaving

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Garcia Tejedor, MDPhD, Principal Investigator — Hospital de Bellvitge. Instituto de Investigación Biomédica de Bellvitge (IDIBELL)
Locations (1):
- Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No